CLINICAL TRIAL: NCT03934853
Title: Human Clinical Study to Confirm Accuracy and Safety of the Inliant Surgical Navigation System for Dental Implant Placement
Brief Title: Study to Confirm Accuracy and Safety of the Inliant Surgical Navigation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navigate Surgical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL-VAV-00862
Record Dates: First submitted 2019-04-11; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Partial Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No arm (Other): There is no arm for this study.
  Interventions: Device: Dynamic Dental Navigation

INTERVENTIONS:
Device: Dynamic Dental Navigation — Aid in dental implant placement in humans

SUMMARY:
A confirmatory dual-clinic, non-randomized study of the Inliant device to aid in dental implant placement in humans. The hypothesis is that using the Inliant Surgical Navigation System ("Inliant") will provide a high degree of accuracy in multiple dimensions relative to the ideal implant position as determined in the planning stage, and will not result in any adverse outcomes related to use of the device. Five clinicians (Investigators) of various clinical backgrounds and experience will use the Inliant device, a licensed, medical device in Canada, to place a dental implant in a total of twenty (20) subjects.

DETAILED DESCRIPTION:
The long term success of dental implant therapy is largely dependent on proper implant positioning in bone, and the facilitation of a well-functioning prosthesis. Surgical complications from implant placement in an incorrect location can include damage to adjacent teeth, sinus perforations, hemorrhage, buccal plate dehiscence, and nerve damage. In implant therapy, dynamic surgical guidance is a new technology used to facilitate accurate and efficient implant placement, and to aid in communication between the restorative dentist and surgeon.

The Inliant device is a dynamic surgical navigation system that is based on passive optical tracking technology. Passive optical tracking is accomplished by having the patient wear a reference body that is identified by an optical tracking system. This information allows the clinician to visualize the surgical drill projected onto a screen, showing its position in 3 dimensions on a CBCT scan of the patient. Dynamic surgical guidance has additional advantages over traditional methods in that it allows for intra-operative changes in implant planning, and allows the clinician to visualize the position of the surgical drill during the procedure.

The purpose of the present study is to analyze the accuracy of the Inliant device as a method of placing dental implants in an actual clinical setting and to confirm its safety.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form (ICF)
* Willing to comply with all study procedures and be available for the study
* Male or female, 22 years of age and older
* In good general health as evidenced by medical history
* To provide attachment of the stent for each implant, there must be at least two adjacent zero mobility teeth anywhere in the same arch on which the surgery is to be performed

Exclusion Criteria:

* A medical condition, psychological condition or dental condition that would exclude a patient from having dental implant surgery. Example: inability to tolerate local anesthesia or other dental disease conditions that would preclude dental implant surgery.
* Use of disallowed concomitant medications (only if a contraindication to dental implant surgery. Examples include long term bisphosphonates, high dose blood thinners, etc.).
* Pregnancy
* Treatment with another investigational drug or other intervention
* Inability to obtain a suitable pre-operative CBCT scan
* In surgery, if there are clinical conditions that unexpectedly do not allow for the placement of an implant, e.g. lack of primary stability during immediate placement.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of implant placement | +/- 7 days of implant procedure
  Uses passive optical tracking technology pre-operatively to plan dental implant placement. Uses the same technology post-operatively for placement comparison assessment.

SECONDARY OUTCOMES:
Safety assessment through collection of adverse event data | +/- 7 days of implant procedure
  Assessment of safety in a clinical environment as determined by review of adverse events related to the use of the device

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas M Makhoul, Principal Investigator — McGill University
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada